CLINICAL TRIAL: NCT06439901
Title: Optimizing the Implementation of Bronchopulmonary Cancer Screening in the Ile de France Region (OPTI-DEPIST-MUT)
Brief Title: Optimizing Bronchopulmonary Cancer Screening
Acronym: OPTI-DEPIST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Collaborators: Institut Mutualiste Montsouris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IC 2023-11
Record Dates: First submitted 2024-05-28; First posted 2024-06-03 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Bronchopulmonary Disease; Diagnoses Disease
Keywords: bronchopulmonary cancer; screening; primary prevention
MeSH Terms: interventions — Mass Screening

STUDY DESIGN:
Intervention Model Description: Multicentre, Interregional , feasibility study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Screening for primary prevention of bronchopulmonary cancer (Other): Screening CTscan according to the NELSON trial schedule (at inclusion, 1 year, 3 years, 5.5 years),
  Interventions: Other: Screening; Other: Inclusion; Other: Chest CTscan and follow-up

INTERVENTIONS:
Other: Screening — A first step to identify and recruit people eligible for screening,
Other: Inclusion — A second step for inclusion of participants, with an online self-questionnaire and information, and an inclusion visit to the health center,
Other: Chest CTscan and follow-up — A third step with an initial CTscan, with dual interpretation and appropriate management of participants, including follow-up care.

SUMMARY:
The aim of this study is to evaluate the feasibility of performing a first screening for bronchopulmonary cancer by thoracic scanner in a French cohort within a dedicated, effective and structured network in the pilot centers participating in the study.

DETAILED DESCRIPTION:
The organization of bronchopulmonary cancer screening in the Ile de France region, within the Mutualists and its affiliated health centers, is based on a clear, simple and functional process:

* Definition of eligibility criteria for screening, based on those of the NELSON study,
* Referral and consultation by a health center physician trained in these criteria,
* Referral and performance of a chest Computer Tomography Scanner (CTscan) according to the same recommendations,
* Structured centralized reading and interpretation of CTscan images,
* Referral to a multidisciplinary team (CITT), if bronchopulmonary cancer is suspected,
* Referral to a tobacco unit in a health center for smokers who have not stopped smoking,
* Organization of follow-up and continuation of the screening program.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged 50 to 74.
* Resident in the Île-de-France region.
* Active smoker or quit smoker for 10 years or less:

  1. more than 10 cigarettes a day for more than 30 years,
  2. more than 15 cigarettes a day for more than 25 years.
* The participant has been informed and has signed the consent form.
* Social Security System affiliation.
* Willingness to participate in a smoking cessation program, if currently smoking.

Exclusion Criteria:

* Active cancer or a history of cancer in remission for less than 5 years (except basal cell carcinoma of th skin or epithelioma in situ of the uterine cervix).
* Presence of symptoms suggestive of bronchopulmonary cancer. Participants with these symptoms require immediate diagnostic investigations and are therefore not eligible for screening.
* Weight >= 140 kg.
* Severe comorbidity contraindicating therapeutic options or invasive thoracic diagnostic investigations.
* Inability to climb two flights of stairs without stopping.
* A thoracic CTscan performed within the previous year.
* Persons deprived of liberty or under guardianship.
* Impossibility to undergo the medical monitoring of the trial for geographical, social or psychological reasons.

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-01-17 (Actual); Primary Completion 2032-01-17 (Estimated); Study Completion 2033-01-17 (Estimated)

PRIMARY OUTCOMES:
Rate of first CTscan for bronchopulmonary cancer screening | 36 months
  Rate of completion of a first bronchopulmonary cancer screening among people who have joined the program (i.e. registered on the program's web platform and met the inclusion criteria).

SECONDARY OUTCOMES:
Eligibility rate among people registering on the web platform | 36 months
  Ratio of the number of eligible people (meeting all inclusion and inclusion criteria and no non-inclusion criteria) to the total number of people registered on the web platform.
Rate of completion of the inclusion visit among people registered on the web platform, | 36 months
  Ratio of the number of people who have completed the inclusion visit to the total number of eligible people registered on the web platform
Rate of completion of screening scanners at 1 year according to NELSON trial schedule | 48 months
  Ratio of the number of people who had their 1-year screening CTscan among those eligible for a 1-year CTscan
Rate of completion of screening scanners at 3 years according to NELSON trial schedule | 72 months
  Ratio of the number of people who had their 3-year screening CTscan among those eligible for a 3-year CTscan
Rate of completion of screening scanners at 5.5 years according to NELSON trial schedule | 102 months
  Ratio of the number of people who had their 5.5-year screening CTscan among those eligible for a 5.5-year CTscan
Correlation of demographic characteristics and the detection of a nodule during the 4 CTscan | 102 months
  Demographic characteristics at inclusion will be compared between people who have or have not had at least one nodule detected on one of the 4 CTscan.
Rate of complications related to complementary explorations | 102 months
  Ratio between the number of people with complications related to complementary explorations and the population having undergone a CT scan.
Smoking cessation rates during the screening program | 102 months
  The rate of newly non-smoking subjects will be calculated for each type of approach by dividing the number of newly non-smoking subjects by the number of subjects people included in the study.
Rate of early-stage bronchopulmonary cancers identified | 102 months
  Number of bronchopulmonary cancers detected at an early stage (stage I or stage II) to the total number of people who underwent a CTscan at inclusion
Rate of positive screening without bronchopulmonary cancer | 102 months
  The rate of false-positive screening will be calculated by people who have at least one positive screening scanner, but whose histology has not confirmed their malignancy, to the number people who had a scanner

CONTACTS AND LOCATIONS:
Overall Officials: Catherine DANIEL, MD, Study Director — Institut Curie
Locations (8):
- France (8):
  - Centre CTPS Bobigny Bondy, Bobigny
  - Centre Municipal de Santé Simone Veil, Issy-les-Moulineaux
  - Centre Municipal de Santé Jacqueline Akoun-Cornet, Malakoff
  - Centre Municipal de Santé Maurice Ténine, Malakoff
  - Centre de Santé Square de la Mutualité, Paris
  - Institut Curie, Paris
  - Institut Mutualiste Montsouris, Paris
  - Centre de Santé MGEN, Paris

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).